CLINICAL TRIAL: NCT04432428
Title: Safety and Efficacy of Patient Controlled Analgesia Using the Sublingual Sufentanil Tablet System (SSTS) in a Fast Track Rehabilitation Program After Total Knee Arthroplasty
Acronym: Zalviso
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/1741
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain
Keywords: knee surgery; Patient Controlled Analgesia (PCA); Enhansed Recovery After Surgery (ERAS)
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Multicentric interventional prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sufentanil sublingual tablet (Experimental): sufentanil sublingual 15µg tablets
  Interventions: Drug: Sufentanil Sublingual Tablet

INTERVENTIONS:
Drug: Sufentanil Sublingual Tablet — all patients will receive tablets for sublingual use, containing 15 microgram of sufentanil. The sufentanil tablets come in a cartridge (40 tablets) and are administered with a special patient-controlled device that uses thumb tag recognition.
  max dose per hour : 3 tablets of 15µg sufentanil

SUMMARY:
The sufentanil sublingual tablet system (SSTS) is an innovative patient-controlled analgesia (PCA) device for the management of acute moderate to severe postoperative pain in hospital settings in adult patients.

The SSTS is non-invasive and imposes no restrictions on patient mobility, which renders it particularly suitable for clinical conditions where early mobilization is a key component of successful surgical outcome.

The present study tests the hypothesis that SSTS is an efficient and safe analgesic technique allowing fast track rehabilitation after total knee arthroplasty in a prospective cohort design.

DETAILED DESCRIPTION:
Total knee arthroplasty is one of the most common major procedures performed today with a significant impact on health care budgets. Fast track rehabilitation programmes are being developed to control hospitalization costs associated with this procedure. Interestingly, such pathway controlled fast track programs also appear to enhance functional recovery and to reduce complications. These beneficial effects are mainly attributed to the practice of rapid mobilization and early intensified physiotherapy which can only be achieved with effective analgesic techniques.

Current PCA techniques - predominantly morphine based - are the gold standard for this purpose but they involve intravenous access and a programmable computer system requiring close supervision. Reported shortcomings are systems failure leading to analgesic gaps, drug errors and restrictions in mobility since patients are tethered to IV poles. The SSTS may overcome these limitations because the opioid used, sufentanil, has a more predictable time of onset, the delivery system does not require programming, and the device does not limit patient's mobility. It retains the benefits of potent analgesia as well as patient empowerment and is particularly suited to target the analgesic effect precisely to the level required in physiotherapeutic sessions.

The present study will test the hypothesis that SSTS is an efficient and safe analgesic technique allowing fast track rehabilitation after total knee arthroplasty in a prospective cohort design.

The study will focus on the efficiency of STSS which is defined as 75% or more of the treated patients proves NRS score less than 4 during 48 hours postoperatively, additionally to the basic pain treatment (paracetamol and NSAID).

The STSS will allow the patient tot take a maximum of 3 doses in one hour. Treatment with the STSS is continued over a period of 48 hours or if necessary up to 72 hours.

During this period the patients pain en parameters will be monitored closely.

The maximum administered total dose of Zalviso will not exceed 1.2mg.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 40-75 years old
* Able to give consent
* Scheduled of elective knee arthroplasty with a fast rehabilitation program
* Able to understand PCA principle and capable to operate SSTS device

Exclusion Criteria:

* Outside age range
* Contra indication for anti-inflammatory drugs
* Revision total knee arthroplasty
* history of substance abuse,
* pregnancy,lactation
* severe hepatic impairment (INR>1,5 and/or AST/ALT above x3 highest normal value),
* sleep apnea (documented by sleep laboratory study),
* severe chronic kidney disease (eGFR<30 mL/min/1.73 m2),
* severe and very severe COPD (GOLD III and IV)
* opioid tolerance (use of >15mg oral morphine equivalent per day within the past 3 months),
* chronic pain conditions necessitating gabapentinoids, steroids or anti-inflammatory drugs
* hypersensitivity to sufentanil
* significant respiratory depression (need for outpatient supplemental oxygen therapy),
* participation in another clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Total time NRS<4 | from end of surgery until 48 hours postoperatively
  cumulative time that patient had NRS<4

SECONDARY OUTCOMES:
length of hospital stay | from hospital admission until hospital discharge, up to 1 week post-operatively
  amount of days that patient was admitted to the hosptial
Incidence of the side effect nausea | from end of surgery until 72 hours postoperatively
  Incidence of the side effect nausea with a simple scale (none, mild, moderate, severe)
Incidence of the side effect vomiting | from end of surgery until 72 hours postoperatively
  Incidence of the side effect vomiting with a simple scale (none, mild, moderate, severe)
Incidence of the side effect itching | from end of surgery until 72 hours postoperatively
  Incidence of the side effect itching with a simple scale (none, mild, moderate, severe)
Incidence of the side effect drowsiness | from end of surgery until 72 hours postoperatively
  Incidence of the side effect drowsiness with a simple scale (none, mild, moderate, severe)
Incidence of the side effect constipation | from end of surgery until 72 hours postoperatively
  Incidence of the side effect constipation with a simple scale (none, mild, moderate, severe)
Oxygen desaturation | from end of surgery until 72 hours postoperatively
  Oxygen desaturation
patient satisfaction with Zalviso PCA | after discontinuation of study medication, up to 72 hrs after start of the study medication
  patient satisfaction assessed with patient ease of care questionnaire
health care worker satisfaction with the patients pain treatment with Zalviso PCA | after patients discontinuation of study medication, up to 1 week after stop study medication
  health care worker satisfaction assessed with nurse/physical therapist ease of care questionnaire
consumption of study medication | from start administration of study medication until end of administration of study medication, up to a maximum of 72 hrs
  total amount of study medication that was administered
Level of analgesia during physiotherapy | from start until end of physiotherapy session, up to 2 days post-operatively
  Level of analgesia during physiotherapy assessed with NRS scale

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wouters, MD PhD, Principal Investigator — University Hospital, Ghent; Luc Verbacnk, MD, Principal Investigator — Yperman Hospital
Locations (1):
- University Hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No